CLINICAL TRIAL: NCT00120380
Title: Combination Therapy of Bosentan and Aerosolized Iloprost in Idiopathic Pulmonary Arterial Hypertension
Brief Title: Combination Therapy of Bosentan and Aerosolized Iloprost in Idiopathic Pulmonary Arterial Hypertension (IPAH)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Futility analysis
Sponsor: Hannover Medical School (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COMBI
Record Dates: First submitted 2005-07-11; First posted 2005-07-18 (Estimated); Last update posted 2012-08-21 (Estimated); Status verified 2006-01

CONDITIONS: Hypertension
Keywords: Idiopathic pulmonary arterial hypertension
MeSH Terms: conditions — Hypertension; Familial Primary Pulmonary Hypertension

ARMS (2):
- Aerosolized Iloprost (Active Comparator)
  Interventions: Drug: Aerosolized iloprost
- Bosentan monotherapy (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aerosolized iloprost
  Arms: Aerosolized Iloprost
Drug: Placebo
  Arms: Bosentan monotherapy

SUMMARY:
The purpose of this study is to test whether the addition of inhaled iloprost is safe and effective in patients with idiopathic pulmonary arterial hypertension who are already being treated with the endothelin receptor antagonist bosentan.

ELIGIBILITY:
Inclusion Criteria:

* IPAH
* > 3 months treatment with bosentan
* 6 minute walk distance 150 - 425 m

Exclusion Criteria:

* other forms of pulmonary hypertension
* severe comorbidities
* cotreatment with sildenafil or investigational drugs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2004-09; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
6 minute walk test

CONTACTS AND LOCATIONS:
Overall Officials: Marius M Hoeper, MD, Study Chair — Hannover Medical School
Locations (1):
- Hannover Medical School, Hanover, Germany

REFERENCES:
- [Result] Hoeper MM, Leuchte H, Halank M, Wilkens H, Meyer FJ, Seyfarth HJ, Wensel R, Ripken F, Bremer H, Kluge S, Hoeffken G, Behr J. Combining inhaled iloprost with bosentan in patients with idiopathic pulmonary arterial hypertension. Eur Respir J. 2006 Oct;28(4):691-4. doi: 10.1183/09031936.06.00057906. PMID 17012628